CLINICAL TRIAL: NCT06186804
Title: A Multicenter, Single-arm, Open-label, Phase II Clinical Study. This Study Consisting of Part A and Part B to Evaluate the Efficacy and Safety of ABSK021 (Pimicotinib) in Patients With Chronic Graft Versus Host Disease
Brief Title: A Phase II Study Evaluating the Efficacy and Safety of ABSK021 (Pimicotinib)) in the Treatment of cGvHD Chronic Graft Versus Host Disease (cGvHD)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK021-201
Record Dates: First submitted 2023-11-28; First posted 2024-01-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-10

CONDITIONS: cGvHD

STUDY DESIGN:
Intervention Model Description: Patients will be instructed to take a specified dose of ABSK021 at the same time each day. In Cycle 1, the patient should take one dose every morning after waking up; After the 15th day of the 1st cycle, the specified dose may be taken in the morning or evening, but should be taken at the same time every day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABSK021 (Experimental): Patients will be instructed to take a specified dose of ABSK021 at the same time each day.
  Interventions: Drug: ABSK021

INTERVENTIONS:
Drug: ABSK021 — Patients in each phase and dose group will receive continuous treatment with oral administration once a day for 28 days/cycle until conditions for treatment termination are met.

SUMMARY:
This is a multicenter, single arm, open label phase II clinical study in China. This study will evaluate the efficacy and safety of ABSK021 (Pimicotinib) in the treatment of patients with cGvHD who failed first-line therapy.

DETAILED DESCRIPTION:
This is a phase II, open-label study to evaluate safety, tolerability, pharmacokinetics (PK), and clinical benefit of ABSK021 in patients with hormone refractory or relapsed cGvHD. This study consisted of Part A and Part B, all cGvHD patients in this study will receive continuous oral treatment with ABSK021 once a day (QD) in a 28-day cycle, complete the core treatment period and extended treatment period, and receive regular follow-up until the termination of treatment is determined.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent and agree to comply with the requirements and restrictions set out in the informed consent.
2. At the time of signing the informed consent., the patient must be at least 18 years old, regardless of gender ；
3. Allogeneic hematopoietic stem cell transplantation from any donor source using bone marrow, peripheral blood stem cells, or cord blood.
4. Patients who have received at least 1 line of systemic therapy
5. If the patient is being treated with glucocorticoids or calcineurin inhibitor(CNI), the patient should have received a stable dose of the above treatment for not less than 2 weeks prior to the first use of ABSK021.
6. ECOG (Eastern Cooperative Oncology Group Performance Status) physical strength score 0-2;7. The patient had sufficient organ and bone marrow function within 14 days prior to the first use of ABSK021.

8. For patients with Part A only: antifungal drugs that are currently being used in combination with CYP3A4 potent inhibitors should have been continuously used in accordance with regulations for no less than one week before the first use of ABSK021

Exclusion Criteria:

1. In previous treatment, he received highly selective colony stimulating factor 1 receptor (CSF-1R) targeted therapy, including small molecule or large molecule drugs;
2. A known history of allergy to components of the investigational drug composition ;
3. Patients continued to use CYP3A4 in combination with antifungal agents or in the two weeks prior to the initial administration of ABSK021 Strong inducer;
4. The patient has received more than 5 lines of systemic therapy for cGvHD;
5. The patient presented with aGvHD symptoms without cGvHD symptoms ;
6. Any evidence of potential tumor or recurrence of post-transplant lymphoproliferative disease at the screening stage .
7. There are factors that have been determined by the investigators to have a significant influence on oral drug absorption
8. Present with cholestatic disease, or unresolved hepatic sinus obstruction syndrome/venous obstructive disease;
9. active infection.
10. During the screening period, the investigators judged that the patients had insufficient pulmonary function reserve, with FEV1≤ 39% or pulmonary function classification score of 3;
11. Prior treatment (adverse events did not return to ≤ Grade 2 (CTCAE v5.0);
12. Pregnant or lactating women;
13. Patients who are unable to or disagree with contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) at each dose can assess the incidence of DLT in patients during the observation period of DLT (Part A only) | Starting from the first medication, observe for 31 days
  Number of Participants With Adverse Event (AE), Serious Adverse Event, (SAE) and Laboratory Abnormalities Defined as Dose Limiting Toxicities (DLT);
Overall response rate after 6 cycles of treatment | 6 months
  Proportion of participants with CR or PR after 6 cycles of treatment as defined by the 2014 NIH Consensus Development Project on Criteria in cGVHD

SECONDARY OUTCOMES:
Adverse Events | Through study completion, an average of 2 years
  Safety assessments will be carried out during the trial.

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of the Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial Peoplep's Hospital, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Zhujiang, Guangdong
  - Tongji Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - The Fir St Affiliated Hospital,Zhejiang Univer Sity School of Medicine, Hangzhou, Jiangsu
  - The First affiliated hospital of SuZhou University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Teaching Hospital of Xinjiang Medical University, Xinjiang, Xinjiang